CLINICAL TRIAL: NCT01981122
Title: A Randomized, Open-label, Phase 2 Study of Sipuleucel-T With Concurrent Versus Sequential Administration of Enzalutamide in Men With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: A Study of Sipuleucel-T With Administration of Enzalutamide in Men With Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P12-2
Record Dates: First submitted 2013-10-29; First posted 2013-11-11 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent Arm (Experimental): Subjects will receive sipuleucel-T concurrently with enzalutamide (160 mg orally once daily). Enzalutamide treatment will start 2 weeks prior to the first leukapheresis and continue for 52 weeks or until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Biological: sipuleucel-T; Drug: enzalutamide
- Sequential Arm (Experimental): Subjects will receive sipuleucel-T followed by enzalutamide (160 mg orally once daily). Enzalutamide treatment will start approximately 10 weeks after the first infusion of sipuleucel-T and continue for 52 weeks or until disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Biological: sipuleucel-T; Drug: enzalutamide

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Other Names: PROVENGE(R); APC8015
Drug: enzalutamide — Enzalutamide is an androgen receptor inhibitor. It is indicated for the treatment of patients with mCRPC who have previously received docetaxel. The enzalutamide dose used in this study will be 160 mg orally once daily.
  Other Names: Xtandi

SUMMARY:
This is a randomized, open-label study designed to assess the effects of sipuleucel-T when administered concurrently or sequentially with enzalutamide.

DETAILED DESCRIPTION:
This is a randomized, open-label study designed to assess the effects of sipuleucel-T when administered concurrently or sequentially with enzalutamide. This study consists of 3 phases. The screening phase will begin at the completion of the informed consent process and continue through registration. The active phase will begin at registration and continue through the post-treatment visit (30 to 37 days following the last study treatment). The long term follow-up (LTFU) phase will begin after the post-treatment visit and will continue until the subject's death or until Dendreon terminates the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided prior to the initiation of study procedures.
* Age ≥ 18 years.
* Histologically documented adenocarcinoma prostate cancer confirmed by a pathology report from prostate biopsy or a radical prostatectomy specimen.
* Metastatic disease as evidenced by bone metastasis or lymph node metastasis.
* Castrate-resistant prostate cancer as demonstrated by one of the following:

  * Prostate specific antigen progression.
  * Progression of measurable disease.
  * Progression of non-measurable disease by soft tissue disease or bone disease.
* Castration levels of testosterone (≤ 50 ng/dL) achieved via medical or surgical castration.
* Serum PSA (Prostate specific antigen) ≥ 2.0 ng/mL.
* Screening ECOG (The Eastern Cooperative Oncology Group )performance status ≤ 1
* Adequate screening hematologic, renal, and liver function as evidenced by laboratory test results obtained ≤ 28 days prior to registration.
* Negative serology test for human immunodeficiency virus 1 and 2.
* Resides within driving distance (round trip within 1 day) of the clinical trial site for the duration of the active phase.

Exclusion Criteria:

* The presence of known lung, liver, or brain metastases, malignant pleural effusions, or malignant ascites.
* Spinal cord compression, imminent long bone fracture, or any other condition that is likely to require radiation therapy and/or steroids for pain control during the active phase.
* History of stage 3 or greater cancer, excluding prostate cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease free at the time of registration. Subjects with a history of stage 1 or 2 cancer must have been adequately treated and been disease free for ≥ 3 years at the time of registration.
* History of seizures or of predisposing factors for seizures.
* Child-Pugh Class C hepatic insufficiency.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sipuleucel-T, GM-CSF or granulocyte colony stimulating factor (G-CSF).
* Previous treatment with sipuleucel-T or enrollment in a sipuleucel-T trial, regardless of whether the subject received sipuleucel-T or control.
* Previous treatment with enzalutamide.
* Previous treatment with abiraterone acetate.
* Previous treatment with ipilimumab.
* Previous treatment with ketoconazole other than topical use or for treatment of infections (e.g., oral thrush); most recent use must have been ≥ 7 days prior to registration.
* Previous treatment with any immunotherapy or investigational vaccine.
* A requirement for ongoing systemic immunosuppressive therapy. Use of inhaled, intranasal, intra-articular, and topical steroids is allowed. Oral or IV steroids to prevent or treat IV contrast reactions are allowed.
* Previous treatment with chemotherapy for mCRPC, or chemotherapy for any reason ≤ 2 years prior to registration.
* Use of concomitant medications that may lower the seizure threshold or the use of antiseizure medications ≤ 1 year prior to registration.
* Received GM-CSF or G-CSF ≤ 90 days prior to registration.
* Ongoing non-steroidal antiandrogen withdrawal response.
* Any of the following medications or interventions ≤ 28 days prior to registration:

  * Radiation therapy, either via external beam or brachytherapy.
  * Any systemic steroid. Use of inhaled, intra-nasal, intra-articular, and topical steroids is allowed. Oral or IV steroids to prevent or treat IV contrast reactions are allowed.
  * Any systemic therapy for prostate cancer, except for ADT (Androgen deprivation therapy).
  * Any investigational product for prostate cancer.
  * Major surgery requiring general anesthesia, with the exception of placement of central venous catheters.
  * Inducers and inhibitors of cytochrome P450 (CYP) enzyme CYP2C8 (gemfibrozil and rifampin).
  * Medications that are metabolized by CYP3A4, CYP2C9, or CYP2C19 that have a narrow therapeutic index.
  * Inducers of CYP3A4 (including but not limited to phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, and phenobarbital).
* A requirement for treatment with opioid analgesics for cancer-related pain ≤ 21 days prior to registration.
* An active infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5˚ F or 38.1˚ C) ≤ 1 week prior to registration.
* Any medical intervention, any other condition, or any other circumstance which could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown, MD, Study Director — Dendreon Pharmaceuticals, LLC
Locations (19):
- United States (19):
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - The Urology Center of Colorado, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - H. Lee Moffitt Cancer and Research Center, Tampa, Florida
  - Uro Partners/ RMD Clinical Research, Melrose Park, Illinois
  - Fort Wayne Medical Oncology and Hematology, Lutheran Hospital, Parkview Regional Medical Center, Fort Wayne, Indiana
  - Johns Hopkins Medicine - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - GU Research Network, Omaha, Nebraska
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Raleigh Hematology Oncology Associates, D.B.A. Cancer Centers of North Carolina, Raleigh, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, PC, Nashville, Tennessee
  - Urology of Virginia, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Virginia Mason Hospital, Seattle, Washington
  - Northwest Medical Specialties, Rainier Physicians, Tacoma, Washington

REFERENCES:
- [Derived] Antonarakis ES, Subudhi SK, Pieczonka CM, Karsh LI, Quinn DI, Hafron JM, Wilfehrt HM, Harmon M, Sheikh NA, Shore ND, Petrylak DP. Combination Treatment with Sipuleucel-T and Abiraterone Acetate or Enzalutamide for Metastatic Castration-Resistant Prostate Cancer: STAMP and STRIDE Trials. Clin Cancer Res. 2023 Jul 5;29(13):2426-2434. doi: 10.1158/1078-0432.CCR-22-3832. PMID 37058234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Concurrent Arm | Sequential Arm
Started | 25 | 27
Completed | 11 | 7
Not Completed | 14 | 20
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Investigator Or Dendreon Discretion | 0 | 1
Not completed — Death | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concurrent Arm | Sequential Arm | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 15 | 23 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (10.6) | 73.3 (9.0) | 70.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 27 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 27 | 52
Height [Mean (Standard Deviation); unit: Centimeters] | 177.0 (8.0) | 177.2 (6.0) | 177.1 (6.9)
Weight [Mean (Standard Deviation); unit: Kg] | 94.6 (19.4) | 91.2 (13.9) | 92.8 (16.6)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 30.3 (5.1) | 29.0 (4.2) | 29.6 (4.6)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions | 22 | 19 | 41
    ECOG 1=Restricted Strenuous Activity | 3 | 8 | 11
Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤6 | 1 | 2 | 3
    Gleason Score 7 | 4 | 8 | 12
    Gleason Score ≥8 | 19 | 16 | 35
    Missing | 1 | 1 | 2
Time from Diagnosis to Randomization [Mean (Standard Deviation); unit: Years] | 5.1 (5.3) | 6.5 (5.6) | 5.8 (5.5)
Time in Years [Number; unit: years] — Categorical presentation of participants based on time from diagnosis to randomization in this study
  years
    0-5 | 16 | 14 | 30
    6-10 | 5 | 5 | 10
    11-15 | 3 | 6 | 9
    16-20 | 0 | 1 | 1
    21-25 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Peripheral PA2024-specific T Cell Proliferation Response to Sipuleucel-T Over Time Via a T Cell Stimulation Index (SI).
Description: PA2024-specific T cell proliferation responses over time will be compared between the concurrent arm and sequential arm using a repeated measurement mixed model analysis. The unit of analysis for the T cell proliferation data is the stimulation index, defined as the median 3H uptake of 3 wells exposed to antigen divided by the median 3H thymidine uptake of 3 wells exposed to media. The stimulation index will be log-transformed prior to analysis.
Time Frame: Each patient was followed for up to 52 weeks after the first dose of sipuleucel-T. Immune sample draws during the treatment period (Week 0 through Week 4) were to be performed at the patient's pre-leukapheresis visits (Pre-Leuk 2 and Pre-Leuk 3).
Population: Summary of Cellular Proliferation Data Through Week 52. All patients with reported data at a specified time-point were analyzed. Number of patients at each time-point differed across the time-points resulting in patient numbers at each time-point that are not equal to the total number of patients analyzed.
Measure: Mean (Standard Deviation); unit: 10^3 cells/mL
Arm/Group | Concurrent Arm | Sequential Arm
Number analyzed (Participants) | 23 | 26
10^3 cells/mL
  PA2024 Baseline: number analyzed (Participants) | 23 | 25
  PA2024 Baseline | 2.48 (4.76) | 1.48 (.92)
  PA2024 Pre-leuk 2: number analyzed (Participants) | 21 | 26
  PA2024 Pre-leuk 2 | 8.76 (13.40) | 5.08 (7.07)
  PA2024 Pre-leuk 3: number analyzed (Participants) | 21 | 25
  PA2024 Pre-leuk 3 | 23.33 (16.98) | 13.96 (11.90)
  PA2024 Week 6: number analyzed (Participants) | 22 | 18
  PA2024 Week 6 | 17.36 (14.39) | 12.72 (11.83)
  PA2024 Week 10: number analyzed (Participants) | 21 | 21
  PA2024 Week 10 | 15.48 (9.53) | 10.90 (9.07)
  PA2024 Week 14: number analyzed (Participants) | 22 | 21
  PA2024 Week 14 | 17.05 (18.72) | 13.05 (13.28)
  PA2024 Week 20: number analyzed (Participants) | 21 | 18
  PA2024 Week 20 | 22.33 (20.23) | 17.83 (13.80)
  PA2024 Week 26: number analyzed (Participants) | 15 | 18
  PA2024 Week 26 | 27.07 (18.26) | 15.39 (10.58)
  PA2024 Week 40: number analyzed (Participants) | 11 | 10
  PA2024 Week 40 | 18.64 (15.48) | 13.70 (11.28)
  PA2024 Week 52: number analyzed (Participants) | 9 | 7
  PA2024 Week 52 | 16.67 (13.13) | 25.43 (18.72)
Statistical Analysis 1: Comparison: Concurrent Arm vs Sequential Arm; Test type: Superiority; p = .095, Mixed Models Analysis; Repeated Measures

ADVERSE EVENTS:
Time Frame: All SAEs reported or observed during or following the first infusion through 60 days post final infusion were recorded in subject's medical record and reported on an electronic case report form (eCRF). Data collection continued until every subject had been followed for minimum 3 years, had died, or had otherwise gone off study.
Arm/Group | Concurrent Arm | Sequential Arm
All-Cause Mortality (participants affected / at risk) | 14/25 | 15/27
Serious Adverse Events (participants affected / at risk) | 2/25 | 9/27
Other Adverse Events (participants affected / at risk) | 23/25 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Arm (N=25) | Sequential Arm (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis In Device (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 2 (2)
Urinary Incotinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Arm (N=25) | Sequential Arm (N=27)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (4)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous Detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous Floaters (Eye disorders) | 0 (0) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (6)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 7 (10)
Paraesthesis Oral (Gastrointestinal disorders) | 3 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Application Site Rash (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (4)
Chest Discomfort (General disorders) | 0 (0) | 2 (3)
Chest Pain (General disorders) | 1 (1) | 3 (3)
Chills (General disorders) | 2 (4) | 7 (12)
Fatigue (General disorders) | 9 (11) | 17 (19)
Infusion Site Inflammation (General disorders) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 2 (2) | 0 (0)
Injection Site Reaction (General disorders) | 1 (2) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 4 (5)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (4)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 3 (3)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Body Temperature Increased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint Crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hair Follicle Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Seborrhoetic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Altered State of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Coordination Abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 6 (9)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 3 (4) | 5 (6)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder Outlet Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Nocturia (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureteric Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic Obstruction Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oroparyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Cyst Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 3 (3) | 5 (5)
Hypertension (Vascular disorders) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 3 (4) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Coldness (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.

DOCUMENTS (2):
  • Study Protocol (2013-05-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01981122/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT01981122/SAP_001.pdf